CLINICAL TRIAL: NCT07311096
Title: Comparison of the Effectiveness of Interscalene Nerve Block and Serratus Posterior Superior Intercostal Plane Block in Patients Undergoing Arthroscopic Shoulder Surgery
Brief Title: Interscalene Block Versus Serratus Posterior Superior Intercostal Plane Block for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, Omer Doymus, Principal Investigator, Erzurum Regional Training & Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBUERZURUMSHOULDER
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Pain
Keywords: Postoperative pain; Analgesia; Regional Anesthesia; Interscalene brachial plexus block; Serratus posterior superior plane block
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist performing the blocks is aware of the group allocation; all other staff and outcome assessors are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene Brachial Plexus Block (ISB) (Experimental): Patients will receive ISB under ultrasound guidance prior to arthroscopic shoulder surgery using 15 ml 0.25% bupivacaine.
  Interventions: Procedure: Interscalene Brachial Plexus Block (ISB)
- Serratus Posterior Superior Intercostal Plane Block (Experimental): Patients will receive SPSIP block under ultrasound guidance using 30 ml 0.25% bupivacaine
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block (SPSIP)

INTERVENTIONS:
Procedure: Interscalene Brachial Plexus Block (ISB) — Patients receive ultrasound-guided ISB before arthroscopic shoulder surgery. 15 ml of 0.25% bupivacaine is injected using a 22 Gauge 50 mm needle with posterior in-plane approach, targeting C5-C6 roots.
  Arms: Interscalene Brachial Plexus Block (ISB)
Procedure: Serratus Posterior Superior Intercostal Plane Block (SPSIP) — Patients receive ultrasound-guided SPSIP interfascial block in sitting position before surgery. Using a 22 Gauge 10 mm needle, 30 ml of 0.25% bupivacaine is injected between serratus posterior muscle and second rib.
  Arms: Serratus Posterior Superior Intercostal Plane Block

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of interscalene (ISB) and serratus posterior superior intercostal plane block (SPSIP) for postoperative analgesia in patients undergoing elective arthroscopic shoulder surgery. The primary outcome is total 24-hour opioid consumption. Secondary outcomes include pain scores, hemidiaphragmatic paresis incidence and severity, duration of analgesia, and changes in lung function. Participants are randomized into ISB or SPSIP groups; blocks are performed under ultrasound guidance. Postoperative pain is managed with patient controlled analgesia(PCA).

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* The American Society of Anesthesiologists I-III
* Scheduled for elective unilateral arthroscopic shoulder surgery

Exclusion Criteria:

* Refusal to participate in the study
* Allergy to the medications to be used
* History of serious heart, kidney or liver disease
* Neurological deficits or neuropathy
* History of anticoagulant use
* Pre-existing operative respiratory dysfunction
* Having chronic shoulder pain
* Being about to undergo open surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Total 24-Hour Postoperative Opioid Consumption | 0-24 hours postoperatively
  Total intravenous opioid consumption recorded for each patient during the first 24 hours after arthroscopic shoulder surgery, including any rescue analgesia administered.

SECONDARY OUTCOMES:
Incidence and Severity of Hemidiaphragmatic Paresis | Pre-block and 30 minutes post-block
  Ipsilateral hemidiaphragmatic function evaluated by M-mode ultrasonography before block and 30 minutes after block completion. Paresis classified as none (<25% reduction), partial (25-75% reduction), or complete (>75% reduction or paradoxical movement).
Duration of Analgesia | Time interval from block completion to initiation of IV PCA fentanyl in each patient
  0-24 hours post-block
Pulmonary Function Changes (FEV1) | Pre-block and 30 minutes post-block
  Pulmonary function measured with bedside spirometry pre-block and 30 minutes post-block. Forced expiratory volume in 1 second (FEV1) recorded; each measurement performed three times and mean value used.
Pulmonary Function Changes (FVC) | Pre-block and 30 minutes post-block
  Pulmonary function measured with bedside spirometry pre-block and 30 minutes post-block. Forced vital capacity (FVC) recorded; each measurement performed three times and mean value used.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Doymus, MD, Principal Investigator — Erzurum Regional Training & Research Hospital
Locations (1):
- Erzurum Regional Training Research Hospital, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumari P, Kumar A, Aliyar R, Sinha L. Continuous serratus posterior superior intercostal plane block for postoperative analgesia in thoracotomy. Anaesth Crit Care Pain Med. 2025 Sep;44(5):101570. doi: 10.1016/j.accpm.2025.101570. Epub 2025 Jun 14. No abstract available. PMID 40523524
- [Background] Dogan G, Kucuk O, Kayir S, Dal GC, Ciftci B, Zengin M, Alagoz A. Serratus posterior superior intercostal plane block versus thoracic paravertebral block for pain management after video-assisted thoracoscopic surgery: a randomized prospective study. Braz J Anesthesiol. 2025 Sep-Oct;75(5):844647. doi: 10.1016/j.bjane.2025.844647. Epub 2025 Jun 3. PMID 40473018
- [Background] Ozen V, Turan EI, Alver S, Ciftci B, Cakir I, Sahin AS. Serratus Posterior Superior Intercostal Plane Block for Postoperative Analgesia in a Pediatric Patient Undergoing Lobectomy: A Case Report. A A Pract. 2025 May 27;19(5):e01988. doi: 10.1213/XAA.0000000000001988. eCollection 2025 May 1. PMID 40421887